CLINICAL TRIAL: NCT04870437
Title: Impact of ExtraCorporeal Phototherapy (ECP) on Auxiliary Follicular T-lymphocytes and Circulating B-lymphocytes During Chronic AntiBody-Mediated Rejection in Kidney Transplantation: IPECAM
Brief Title: Impact of ExtraCorporeal Phototherapy (ECP) on Auxiliary Follicular T-lymphocytes and Circulating B-lymphocytes During Chronic AntiBody-Mediated Rejection in Kidney Transplantation.
Acronym: IPECAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Therakos (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A00580-41
Record Dates: First submitted 2021-03-30; First posted 2021-05-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Kidney Transplantation
Keywords: Chronic AntiBody-Mediated Rejection; ExtraCorporeal Phototherapy; Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extracorporeal phototherapy (Experimental)
  Interventions: Other: Extracorporeal phototherapy

INTERVENTIONS:
Other: Extracorporeal phototherapy — The principle of ECP is to collect mononucleated cells from the blood by centrifugation. After purification, the mononucleated cells are incubated ex-vivo with a photo-activatable DNA intercalating agent (8-methoxypsoralen, UVADEX®), then re-injected to the patient.

SUMMARY:
Chronic AntiBody-Mediated Rejection (cABMR) is the leading cause of late kidney transplant loss (after 1 year of kidney transplantation). Its therapeutic management is poorly codified and there is currently no treatment referring.

Extracorporeal phototherapy (ECP) is a therapeutic apheresis that involves purifying mononucleated cells in the blood, exposing them to UltraViolet A (UVA) and re-injecting them to the patient. This treatment is used as common care in the first line as part of the treatment of cutaneous T lymphoma and in the second line as part of the graft versus host reaction after bone marrow allograft.

The mechanisms underlying the action of the ECP are not well known. They are mediated by the reinjection of cells exposed to UVA which enter apoptosis and induce immunomodulation. Recent work during cABMR shows that TFH lymphocytes, the maturing population of B lymphocytes, are deregulated and activated.

The hypothesis is that ECP can modulate T Follicular Helper (TFH) lymphocytes during cABMR.

ELIGIBILITY:
Inclusion Criteria:

* ECP treatment decision based on transplant team habits (care management)
* Age ≥ 18 years
* Affiliation to a French social security scheme
* Kidney transplant at least 6 months prior to inclusion
* cABMR proven by a renal graft biopsy less than 3 months and meeting the following histological criteria:

  * allograft glomerulopathy (cg>0, and maximum score cg2) or intimal fibrosis
  * C4d positive or ptc+g greater than or equal to 2
  * Presence of Donor Specific Antibody (DSA)
  * Interstitial Fibrosis and Tubular Atrophy (IFTA) less than or equal to 2
* Glomerular filtration rate > 30 mL/min/1.73 m2
* Signed informed consent to participate in the study

Exclusion Criteria:

* Active infection or infection with hepatitis B, C or HIV virus
* Pregnant, breastfeeding or parturient woman
* Person deprived of liberty by judicial or administrative decision
* Person receiving psychiatric care under duress
* Person subject to legal protection
* Person out of state to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of TFH cells and their activation markers | From the 1st session of ECP to 1 year after the 1st session
  Variation in the frequency of TFH cells and their activation markers under treatment.

SECONDARY OUTCOMES:
Subsequent ECP response in patients with cABMR | 3 months of treatment per ECP
  Study of the 3-month TFH/TFR value of ECP treatment as a marker for subsequent ECP response in patients with cABMR
Concentration of pro and anti-inflammatory cytokines | From the 1st session of ECP to 1 year after the 1st session
  Study of the concentration of pro-inflammatory cytokines (IL-6, TNFα, IL-1β, IL-17, IFN-gamma, IL-21, IL-12, IL-17, CXCL13) and anti-inflammatory cytokines (IL10, TGF-b) over time in ECP
Concentration of circulating B-cell populations | From the 1st session of ECP to 1 year after the 1st session
  Study of the concentration of circulating B-cell populations due to ECP
Measurement of genetic markers in TFH cells | At 1 week of the 1st session of ECP and at 3 month after the 1st session
  Study of genetic markers in TFH cells in cell co-culture in vitro to describe their function
Comparison of clinical data of patients | From the 1st session of ECP to 1 year after the 1st session
  Clinical measures (medical examinations) of patients
Comparison of biological data of patients | From the 1st session of ECP to 1 year after the 1st session
  Biological measures (blood samples) of patients

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Chu Besancon, Besançon
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Chu Saint Etienne, Saint-Etienne
  - CHU de STRASBOURG, Strasbourg

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).